CLINICAL TRIAL: NCT00422877
Title: Phase II Open-Label Study of Weekly Taxoprexin® (DHA-paclitaxel) Injection as Second Line Therapy for Patients With Advanced Primary Cancers of the Liver, Including Hepatocellular Carcinoma and Carcinoma of the Gallbladder or Biliary Tract
Brief Title: Taxoprexin® Treatment for Advanced Primary Cancers of the Liver, Gallbladder or Biliary Tract
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor suspended development of the drug on September 3, 2008.
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P01-05-23
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Last update posted 2025-10-16 (Actual); Status verified 2017-07

CONDITIONS: Cancer of the Liver
Keywords: Liver cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — docosahexaenoyl-paclitaxel; Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Taxoprexin (Experimental): Starting dose of 500 mg/m2 (400 mg/m2 for patients with an elevated bilirubin at baseline) administered intravenously by a 1-hour infusion weekly for the first 5 weeks of a 6 week cycle.
  Interventions: Drug: Taxoprexin

INTERVENTIONS:
Drug: Taxoprexin — Administered by intravenous infusion over 1 hour infusion
  Other Names: Docosahexaenoic acid (DHA)-paclitaxel

SUMMARY:
To evaluate objective response rate and duration of response to weekly Taxoprexin®.

To evaluate the safety profile of weekly Taxoprexin® in this patient population.

To evaluate overall survival in the same patient population.

To evaluate time to disease progression, and the time to treatment failure in patients with primary liver cancer being treated with weekly Taxoprexin® Injection.

To explore the trough and peak blood levels of Taxoprexin® and paclitaxel in these patients.

DETAILED DESCRIPTION:
This is a Phase II open-label study of weekly Taxoprexin® Injection in patients with advanced primary cancers of the liver, including hepatocellular carcinoma (HCC), or carcinoma of the gallbladder or biliary tract (BTC), who have not received prior systemic cytotoxic therapy for advanced disease. Patients may have previously received radiation and/or systemic chemotherapy as adjuvant therapy. Patients may not have been treated previously with a taxane. Patients may have been previously treated with up to two immunological and/or biologic agents (e.g., interferon, monoclonal antibodies, tyrosine kinase inhibitors). Patients will receive Taxoprexin® Injection at a dose of 500mg/m2 (400mg/m2 for patients with an elevated bilirubin at baseline) intravenously by 1-hour infusion weekly for the first five weeks of a six week cycle. Treatment will continue until progression of disease, intolerable toxicity, refusal of continued treatment by patient or Investigator decision.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologic or cytologic confirmation of primary cancer of the liver, including HCC or adenocarcinoma of the gallbladder or bile ducts and advanced (unresectable and/or metastatic) disease.
2. Patients must have at least one measurable lesion by RECIST criteria.
3. Patients may have received up to two prior systemic non-cytotoxic regimens for their disease. Prior treatment with immunologic and/or biologic agents is allowed.
4. At least 6 weeks (42 days) since any prior immunologic or biologic therapy.
5. At least 4 weeks (28 days) since prior radiotherapy to >20% of the bone marrow or prior adjuvant chemotherapy.
6. Lesions being used to assess disease status may not have been radiated or if so, must have progressed during or after radiation therapy.
7. Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
8. Patients must be at least 18 years of age.
9. Patients must have adequate liver and renal function.
10. Patients must have adequate bone marrow function.
11. Patients must sign an informed consent form indicating that they are aware of the investigational nature of this study and in keeping with the policies of the institution.

Exclusion Criteria:

1. Patients who have received prior therapy with any taxane.
2. Patients who have a past or current history of cancer other than the entry diagnosis, except for curatively treated non-melanoma skin cancer or carcinoma in situ of the cervix or other cancers treated for cure and with a disease-free survival longer than 5 years.
3. Patients with symptomatic brain metastasis (es).
4. Patients who are pregnant or nursing and patients who are not practicing an acceptable method of birth control. Patients may not breastfeed while on this study.
5. Patients with active infections currently receiving anti-infectious treatment (e.g., antibiotics, antivirals, or antifungals).
6. Patients with current peripheral neuropathy of any etiology that is greater than grade one (1).
7. Patients with unstable or serious concurrent medical conditions are excluded.
8. Patients with a known hypersensitivity to Cremophor®.
9. Patients with one or more of the following as the only manifestations of disease are ineligible: bone lesions, leptomeningeal disease, ascites, pleural/pericardial effusions, carcinomatous lymphangitis, central nervous system (CNS) metastases, lesions in a previously irradiated area that have not shown definite progression, or disease only inferred from laboratory tests or markers.
10. Patients with a history of Gilbert's Syndrome.
11. Patients must not receive any concurrent chemotherapy, radiotherapy, non-FDA approved nutritional supplements or herbal preparations or immunotherapy while on study.
12. Known HIV disease or infection.
13. Patients receiving ketoconazole, erythromycin, verapamil, diazepam, quinidine or diltiazem.
14. Patients must not have had any surgical procedure requiring hospitalization and administration of general anesthesia within the past 28 days.
15. Patients must not have received prior systemic chemotherapy for advanced disease. Prior adjuvant systematic chemotherapy (non-taxane containing) is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Achieved an Objective Complete Response (CR) or Partial Response (PR) | Assessed every 6 weeks, up to 12 months
  Antitumor response was defined as the percentage of participants who achieved an objective response (Confirmed Response [CR] or Partial Response [PR]), confirmed by repeat assessments performed no less than 4 weeks after the criteria for response were first met. Response was based on the blinded radiological review using Response Evaluation Criteria in Solid Tumors (RECIST) response guidelines, Version 1.0.
  A complete response was defined as a disappearance of all target lesions determined by 2 consecutive observations not less than 4 weeks apart.
  Partial response was defined as a 30% decrease in the sum of the longest diameters (LD) of target lesions, taking as reference the baseline sum of LD determined by 2 consecutive observations not less than 4 weeks apart.

SECONDARY OUTCOMES:
Time to progression (TTP) | Up to 12 months
  TTP was defined as the time from randomization to documented first disease progression. Progressive disease was defined as at least a 20% increase in the sum of longest diameter (LD) of target lesions, taking as references the smallest sum LD recorded since treatment start or the appearance of 1 or more lesions.
Time to Treatment Failure (TTF) | Baseline to stopping treatment
  TTF is defined as the time from randomization to the discontinuation of protocol treatment for any reason
Overall Participant Survival | Up to 12 months
  Overall survival was defined as the time from the day of randomization and ends at either death of the participant or the termination of the study, whichever came first. Participants were followed every 2 months, whether on or off study, for survival information. Participants alive at the time of termination of the study were considered censored.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Kaseb, M.D., Study Director — M.D. Anderson Cancer Center
Locations (1):
- University of Texas, MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No